CLINICAL TRIAL: NCT05755022
Title: Reverse Engineering Utilizing the 3D Photogrammetry Technique Versus Commercial Scanners for Accurate Repositioning of the Maxilla After Le-fort I Osteotomy for Correction of the Dentofacial Deformity (Randomized Controlled Clinical Trial).
Brief Title: 3D Photogrammetry Versus Commercial Scanners for Accurate Repositioning of the Maxilla for Correction of the Dentofacial Deformity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Yacoub Girgis, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-2022-12-10
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Dentofacial Deformities
Keywords: 3D Photogrammetry; Reverse Engineering; Orthognathic Surgery; Pre-bent Plates
MeSH Terms: conditions — Dentofacial Deformities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary segment repositioning by utilizing reverse engineering using the 3D photogrammetry. (Experimental): * The printed stereolithographic model with the adapted miniplates will be scanned using 3D photogrammetry technique and a specific software dedicated for image acquisition will be used.
  * A guide will be designed on the reproduced virtual model. This guide will be used intraoperative as a locating and positioning guide for the maxilla and the plates.
  Interventions: Procedure: Maxillary Segment Repositioning
- Maxillary segment repositioning by utilizing reverse engineering using the commercial scanners. (Active Comparator): • The printed stereolithographic model with the adapted miniplates will be scanned using the commercial scanners and imported for virtual designing of the positioning and locating guide that will be used intraoperative for positioning the maxilla.
  Interventions: Procedure: Maxillary Segment Repositioning

INTERVENTIONS:
Procedure: Maxillary Segment Repositioning — * Le-Fort I osteotomy will be made using the cutting guide.
  * Mobilization of the maxilla will be done.
  * The osteotomized segment will be positioned using the positioning guide that will be fabricated utilizing the reverse engineering technology using 3D photogrammetry technique.
  * While the guide in place, the plates will be fixed into their intended position.
  * After fixation of the plates, the guide will be removed.
  Arms: Maxillary segment repositioning by utilizing reverse engineering using the 3D photogrammetry.
Procedure: Maxillary Segment Repositioning — * Le-Fort I osteotomy will be made using the cutting guide.
  * Mobilization of the maxilla will be done.
  * The osteotomized segment will be positioned using the positioning guide that will be fabricated utilizing the reverse engineering technology using the commercial scanners.
  * While the guide in place, the plates will be fixed into their intended position.
  * After fixation of the plates, the guide will be removed.
  Arms: Maxillary segment repositioning by utilizing reverse engineering using the commercial scanners.

SUMMARY:
Current advances in the three-dimensional virtual surgical planning (3D-VSP) of the orthognathic surgery have brought newer insights, enormous benefits and have become an indispensable aid for diagnosis, treatment planning and outcome assessment especially in the management of dentofacial deformities.

The extent to which the planned surgical outcome could be achieved is dependent on the surgeon's ability to accurately transfer the planned movements to the real surgical field. Accurate repositioning of the maxilla after Le-fort I osteotomy is of utmost importance for an esthetic and functional purposes.

The goal of this interventional study is to compare the 3D photogrammetry technique versus the commercial scanners for accurate repositioning of maxillary segment after le-fort I osteotomy using the reverse engineering technology.

The main question it aims to answer; Is the utilization of the 3D Photogrammetry technique affect the accuracy of maxillary segment repositioning after le-fort I osteotomy compared with the commercial scanners?

DETAILED DESCRIPTION:
In orthognathic surgery, the precise repositioning of the maxilla after Le-fort I osteotomy is a challenging procedure because there is no room for error in this step if the procedure is to be accurate.Transferring the virtual position of the maxilla to the real operative field via the intermediate occlusal splint fabrication, which is the most commonly used method, ensures only the intended position of the maxilla in the transverse, sagittal planes and cannot guarantee its vertical position in relation to the skull base. The vertical maxillary repositioning usually relies on a manual intraoperative adjustment using either intra-oral or extraoral reference points and affected by the degree of autorotation of the mandible that occur as a result of the surgical maneuvers operated by the surgeon intraoperatively. This makes the reliability of and precision in transferring virtual surgical plans to the operative field is still unpredictable defeating the main advantages of 3D technology. Moreover, it can be time consuming.

Many attempts to obtain a more reliable method for positioning the maxilla, independent of the mandible, have been made such as a series of maxillary reposition templates, patient specific osteosynthesis plates and navigation assisted surgery and it yielded satisfactory results. Also, intraoperative occlusal-based devices that transfer virtual surgical planning to the operating field for repositioning of the osteotomized segments was introduced. Most of the time the surgeon looks for new modalities to optimize his surgical results, simplify the execution of the surgery and at the same time to meet the patients' demands and expectations.

Photogrammetry is a versatile, readily available technique that allows for creating a 3D model from 2D photographs in an affordable manner and with a high levels of precision equivalent to other tools that are generally more expensive and less available such as a commercial scanner. It has several applications in the life and earth sciences, medicine, osteological studies, architecture, topography, archaeology, crime scene investigation, cinematography, and engineering. So, the present study aims to assess the accuracy gained and the feasibility of using this technique for transferring the virtually intended maxillary segment position to the real operation compared with the commercial scanners.

Trial design:

Randomized Controlled Clinical Trial. Parallel group, two arm with allocation ratio 1:1.

Sample size:

This study will be conducted for 24 patients, 12 patients per group.

Patients will be selected from the outpatient clinics of Oral and Maxillofacial Surgery Department and Orthodontic Department, Faculty of Dentistry, Cairo University. The trial is to be conducted in the Oral and Maxillofacial Surgery Department, Cairo University.

The eligible patients will be randomly allocated into 2 groups:

Intervention group; Maxillary segment repositioning using positioning guide for the maxilla and the pre-bent plates that is fabricated by the reverse engineering technology utilizing the 3D photogrammetry technique.

Comparator group; Maxillary segment repositioning using positioning guide for the maxilla and the pre-bent plates that is fabricated by the reverse engineering technology utilizing the commercial scanners.

General operative procedures:

Patients of both groups will be subjected to:

* Comprehensive clinical and radiographic examination.
* Pre-operative photographs will be taken.
* Primary upper and lower impressions will be made for the selected patients and the impression material will be poured using hard dental stone to make dental models.

Surgical planning / Preoperative workup;

For both groups:

* Virtual planning: Using dedicated software, 3D digitized bony maxilla will be virtually osteotomized and repositioned to the new intended postoperative position.
* Printing of the corrected 3D model and plate pre-bending (2.0 titanium mini plates will be selected and perfectly adapted over the corrected and printed 3D model).
* Scanning of plate adapted on the printed 3D model to generate a virtual model.

  * For the intervention group; Pre-bent plates will be scanned using 3D photogrammetry technique and a specific software dedicated for image acquisition will be used.
  * For the Comparator group; Pre-bent plates will be scanned using the commercial scanners and imported for virtual designing of the positioning and locating guide.
* A guide will be designed on the reproduced virtual model. This guide will be used intraoperative as a locating and positioning guide for the maxilla and the plates.
* To ensure a more precise location of the positioning guide, the cutting guide will be also constructed and act as a cutting and screw hole locating guide as well. This will be done by incorporating the drill holes to be used for final placement and fixation of the maxilla, in the cutting guide.

Surgical procedure:

* The procedure will be performed under general anesthesia with nasotracheal intubation and controlled hypotension.
* Lidocaine Hydrochloride with 1:200,000 of Epinephrine solution will be utilized for hemostasis.
* Scrubbing and draping of the patient will be carried out in a standard fashion.
* Intra-oral maxillary vestibular incision will be used, elevation of the flap and dissection will be performed exposing the antero-lateral and posterior-lateral aspects of the maxilla.
* Cutting surgical guide will be adapted over the maxilla, the screw holes incorporated in the surgical guide will be drilled and then the osteotomy will be performed and completed using chisels.
* Mobilization of the maxilla will be done. Finally, the positioning and locating guide for the maxilla and the plates will be used. While the guide in place, the plates will be fixed into their position.
* After fixation of the plates, the guide will be removed.
* The rest of the orthognathic surgery (mandibular osteotomy, genioplasty if needed) will be completed in a conventional fashion.
* Debridement, irrigation of the surgical field followed by wound closure and suturing using 3-0 resorbable suture.

Postoperative care:

* Ice packs will be applied for 20 minutes every 1 hour for the first 24 hours to minimize the edema.
* High caloric soft diet will be instructed.
* Good oral hygiene will be emphasized.
* All patients will be kept on the following regimen;

  * Ampicillin/sulbactam 1500 mg vial Intra-muscular( IM) injection every 12 hours for 5 days.
  * Oral Metronidazole 500 mg every 8 hours for 5 days.
  * Diclofenac sodium75 mg IM injection whenever needed.
  * Diclofenac Potassium 50 mg tablets will be given every 8 hours for control of pain.
  * Dexamethasone sodium phosphate 8 mg/2ml IM injection on 8 doses, the first 4 doses will be given every 6 hours, and then it will be tapered on next 4 doses to half the dose every 6 hours.
  * Methylprednisolone acetate 80 mg/ml IM injection will be given with the last dose of Dexamethasone sodium phosphate.
  * The oral antibiotic regimen (Amoxicillin/Clavulanic acid 1000 mg everym12 hours) will be continued for 5-7 days postoperatively to guard against infection.

Number of visits & follow up period:

* All patients will be advised to stay on a soft diet for 4-6 weeks to avoid any undue forces on the surgical site.
* Postoperative CT will be obtained one week postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-60 years.
* Patients requiring one-piece Le-Fort I osteotomy as part of their orthognathic surgery for the correction of dentofacial deformity.
* Patients should be free from any significant medical condition that could affect or hinder normal healing and predictable outcomes.
* Patients with no signs or symptoms of temporomandibular joint disorders.
* Patients who will be committed to the follow up period and agree to sign the informed consent.

Exclusion Criteria:

* Patients requiring segmental Le-Fort I osteotomy.
* Patients with previous history of orthognathic surgery.
* Patients with cleft lip and palate.
* Patients with skeletal deformities owing to trauma or tumor resection.
* Patients with any intra-bony lesions or infections.
* Patients with temporomandibular joint disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of maxillary segment repositioning | Outcome will be assessed with immediate postoperative Computed Tomography at one week.
  The actual postoperative 3D maxillary segment position will be compared with the preoperative virtual maxillary positioning by:
  A) Linear and angular measurements:
  Some specific reproducible points and planes will be identified on the 3D virtual model, and then on the post-surgery model. The distance from points to planes will be calculated on each model and the difference between these distances is to be registered as the error of accuracy.
  B) Color-coded map:
  Different colors show the distance between the surfaces, with green color usually showing the lack of distance, meaning zero error of accuracy. This method of assessing changes in 3D surfaces involves measuring the point-to-point distance of one mesh (VSP - 3D model reference) to the second mesh (Postoperative - 3D model test) and generating a color distance map.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Beheiri, PhD, Study Director — Professor; Samer Noman, PhD, Study Director — Assistant Professor; Sherif A Hassan, PhD, Study Director — Assistant Professor; Dina Y Girgis, Master, Principal Investigator — Assistant lecturer
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Egypt

REFERENCES:
- [Background] Ong TK, Banks RJ, Hildreth AJ. Surgical accuracy in Le Fort I maxillary osteotomies. Br J Oral Maxillofac Surg. 2001 Apr;39(2):96-102. doi: 10.1054/bjom.2000.0577. PMID 11286442
- [Background] Mazzoni S, Bianchi A, Schiariti G, Badiali G, Marchetti C. Computer-aided design and computer-aided manufacturing cutting guides and customized titanium plates are useful in upper maxilla waferless repositioning. J Oral Maxillofac Surg. 2015 Apr;73(4):701-7. doi: 10.1016/j.joms.2014.10.028. Epub 2014 Nov 29. PMID 25622881
- [Background] Pascal E, Majoufre C, Bondaz M, Courtemanche A, Berger M, Bouletreau P. Current status of surgical planning and transfer methods in orthognathic surgery. J Stomatol Oral Maxillofac Surg. 2018 Jun;119(3):245-248. doi: 10.1016/j.jormas.2018.02.001. Epub 2018 Feb 22. PMID 29476926
- [Background] Pietzka S, Mascha F, Winter K, Kammerer PW, Sakkas A, Schramm A, Wilde F. Clinical Accuracy of 3D-Planned Maxillary Positioning Using CAD/CAM-Generated Splints in Combination With Temporary Mandibular Fixation in Bimaxillary Orthognathic Surgery. Craniomaxillofac Trauma Reconstr. 2020 Dec;13(4):290-299. doi: 10.1177/1943387520949348. Epub 2020 Aug 17. PMID 33456700
- [Background] Kraeima J, Schepers RH, Spijkervet FKL, Maal TJJ, Baan F, Witjes MJH, Jansma J. Splintless surgery using patient-specific osteosynthesis in Le Fort I osteotomies: a randomized controlled multi-centre trial. Int J Oral Maxillofac Surg. 2020 Apr;49(4):454-460. doi: 10.1016/j.ijom.2019.08.005. Epub 2019 Sep 8. PMID 31506186
- [Background] Heufelder M, Wilde F, Pietzka S, Mascha F, Winter K, Schramm A, Rana M. Clinical accuracy of waferless maxillary positioning using customized surgical guides and patient specific osteosynthesis in bimaxillary orthognathic surgery. J Craniomaxillofac Surg. 2017 Sep;45(9):1578-1585. doi: 10.1016/j.jcms.2017.06.027. Epub 2017 Jul 8. PMID 28793965
- [Background] Hernandez-Alfaro F, Guijarro-Martinez R. New protocol for three-dimensional surgical planning and CAD/CAM splint generation in orthognathic surgery: an in vitro and in vivo study. Int J Oral Maxillofac Surg. 2013 Dec;42(12):1547-56. doi: 10.1016/j.ijom.2013.03.025. Epub 2013 Jun 13. PMID 23768749
- [Background] Jabar N, Robinson W, Goto TK, Khambay BS. The validity of using surface meshes for evaluation of three-dimensional maxillary and mandibular surgical changes. Int J Oral Maxillofac Surg. 2015 Jul;44(7):914-20. doi: 10.1016/j.ijom.2015.02.005. Epub 2015 Mar 6. PMID 25752242
- See also: Surgical accuracy in Le Fort I maxillary osteotomies — http://pubmed.ncbi.nlm.nih.gov/11286442/
- See also: Computer-aided design and computer-aided manufacturing cutting guides and customized titanium plates are useful in upper maxilla waferless repositioning — http://pubmed.ncbi.nlm.nih.gov/25622881/
- See also: Current status of surgical planning and transfer methods in orthognathic surgery — http://pubmed.ncbi.nlm.nih.gov/29476926/
- See also: Clinical Accuracy of 3D-Planned Maxillary Positioning Using CAD/CAM-Generated Splints in Combination With Temporary Mandibular Fixation in Bimaxillary Orthognathic Surgery — https://pubmed.ncbi.nlm.nih.gov/33456700/
- See also: Splintless surgery using patient-specific osteosynthesis in Le Fort I osteotomies: a randomized controlled multi-centre trial — https://pubmed.ncbi.nlm.nih.gov/31506186/
- See also: Clinical accuracy of waferless maxillary positioning using customized surgical guides and patient specific osteosynthesis in bimaxillary orthognathic surgery — https://pubmed.ncbi.nlm.nih.gov/28793965/
- See also: New protocol for three-dimensional surgical planning and CAD/CAM splint generation in orthognathic surgery: an in vitro and in vivo study — https://pubmed.ncbi.nlm.nih.gov/23768749/
- See also: The validity of using surface meshes for evaluation of three-dimensional maxillary and mandibular surgical changes — https://pubmed.ncbi.nlm.nih.gov/25752242/